CLINICAL TRIAL: NCT03736707
Title: High-Frequency Oscillation Ventilation Versus Conventional Mechanical Ventilation in Very Preterm Infants With Perinatal Acute Respiratory Distress Syndrome: Multicenters Randomized Controlled, Superiority Trial
Acronym: HFOV for ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Jiulongpo No.1 People's Hospital (Other); Chongqing Maternal and Child Health Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Peking University Third Hospital (Other); First Hospital of Tsinghua University (Other); Women and Children's Hospital, Branch of Chongqing Sanxia Central Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Quanzhou Children's Hospital (Other); Xiamen Maternity & Child Care Hospital (Other); Zhujiang Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Academy of Medical Science and General Hospital (Other); Guangdong Women and Children Hospital (Other); Women and Children's Health Hospital of Yulin (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guiyang Maternal and Child Health Care Hospital (Other); The First People's Hospital of Zunyi (Other); Lanzhou University Second Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); LanZhou University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Zhengzhou Children's Hospital, China (Other); Third Affiliated Hospital of Zhengzhou University (Other); the Maternal and Child Health Hospital of Hainan Province (Other); Bethune International Peace Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Children's Hospital of Nanjing Medical University (Other); The First Hospital of Jilin University (Other); Children's Hospital of Fudan University (Other); Maternal and Children's Healthcare Hospital of Taian (Other); The Second Hospital of Shandong University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Chengdu Women and Children's Center Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Affiliated Hospital of Southwest Medical University (Other); Shenzhen People's Hospital, The Second Medical College of Jinan University (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Kunming Children's Hospital (Other); The First People's Hospital of Yunnan (Other); First Affiliated Hospital of Kunming Medical University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Women and Children's Health Hospital of Qujing (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); The First People's Hospital of Yinchuan (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Beijing 302 Hospital (Other); Hunan Children's Hospital (Other Government); Women and Children Hospital of Qinghai Province (Other); Jiangxi Province Children's Hospital (Other); Inner Mongolia People's Hospital (Other); Mianyang Central Hospital (Other); People's Liberation Army No.202 Hospital (Other); Ningbo Women & Children's Hospital (Other); Shanghai Children's Medical Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Nanjing Medical University (Other); Xianyang Children's Hospital (Other); Qinhuangdao Maternal and Child Health Care Hospital (Other); Xuzhou Children Hospital (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Principal Investigator, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFOV for perinatal ARDS; CSTB2024NSCQ-MSX0158 (Other: Natural Science Foundation of Chongqing)
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome; High Frequency Oscillatory Ventilation; Preterm; Conventional Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Intervention Model Description: Very preterm neonates with perinatal acute respiratory distress syndrome will be randomized and assigned to high frequency oscillation ventilation (HFOV) or conventional mechanical ventilation (CMV)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The caregivers will not be blinded, and the outcome assessors and data analysts will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high frenquency oscillation ventilation (HFOV) (Experimental): HFOV + volume guarantee (VG) as the intervention group HFOV was provided only with piston or membrane oscillators capable of delivering true oscillatory pressure with an active expiratory phase (i.e., Acutronic FABIAN-III, SLE 5000, Löwenstein Med LEONI+, or Sensormedics 3100A). Other machines offering high frequency ventilation were excluded. The lung recruitment maneuver was performed as previously described,15 and lung volume was assessed by chest radiography or lung ultrasound, targeting the right diaphragm at the level of 8th-9th rib (or 7th-8th rib in case of air leak).
  Crossover between HFOV and CMV This study allowed infants who failed to respond to their assigned ventilation mode to receive a trial of the alternate mode. Crossover criteria for HFOV-assigned neonates included failure for 3 hours to maintain SpO2 ≥ 50% despite FiO2 of 1.0, PaCO2 > 60 mmHg for 3 hours, or signs of ventilator-induced cardiac output reduction. Non-responders to HFOV were switched to CMV.
  Interventions: Device: HFOV
- conventional mechanical ventilation (CMV) (Active Comparator): CMV was delivered by time-cycled, pressure-limited ventilators. Only pressure regulated volume control (PRVC) will be provided by any type of neonatal ventilator.
  Crossover criteria for CMV-assigned neonates included failure for 3 hours to maintain SpO2 ≥ 50% despite FiO2 of 1.0, PaCO2 > 60 mmHg for 3 hours, or requiring > 30 cm H2O PIP to sustain ventilation. Non-responders to CMV were switched to HFOV.
  in both groups, ventilator settings were adjusted at the discretion of the attending clinician to maintain a SpO2 between 90%-94%, a PaO2 between 50 and 80 mm Hg and a PaCO2 between 35 and 60 mm Hg and a pH between 7.20 and 7.45. PO2 and PCO2 levels were monitored using arterial blood gas analysis and/or transcutaneous monitoring.
  Interventions: Device: CMV

INTERVENTIONS:
Device: HFOV — HFOV + volume guarantee (VG) as the intervention group HFOV was provided only with piston or membrane oscillators capable of delivering true oscillatory pressure with an active expiratory phase (i.e., Acutronic FABIAN-III, SLE 5000, Löwenstein Med LEONI+, or Sensormedics 3100A). Other machines offering high frequency ventilation were excluded. The lung recruitment maneuver was performed as previously described, and lung volume was assessed by chest radiography or lung ultrasound, targeting the right diaphragm at the level of 8th-9th rib (or 7th-8th rib in case of air leak).
  Crossover between HFOV and CMV This study allowed infants who failed to respond to their assigned ventilation mode to receive a trial of the alternate mode. Crossover criteria for HFOV-assigned neonates included failure for 3 hours to maintain SpO2 ≥ 50% despite FiO2 of 1.0, PaCO2 > 60 mmHg for 3 hours, or signs of ventilator-induced cardiac output reduction. Non-responders to HFOV were switched to CMV.
  Arms: high frenquency oscillation ventilation (HFOV)
Device: CMV — CMV as the standard group CMV was delivered by time-cycled, pressure-limited ventilators. Only pressure regulated volume control (PRVC) will be provided by any type of neonatal ventilator.
  Crossover criteria for CMV-assigned neonates included failure for 3 hours to maintain SpO2 ≥ 50% despite FiO2 of 1.0, PaCO2 > 60 mmHg for 3 hours, or requiring > 30 cm H2O PIP to sustain ventilation. Non-responders to CMV were switched to HFOV.
  Ventilator settings were adjusted at the discretion of the attending clinician to maintain a SpO2 between 90%-94%, a PaO2 between 50 and 80 mm Hg and a PaCO2 between 35 and 60 mm Hg and a pH between 7.20 and 7.45. PO2 and PCO2 levels were monitored using arterial blood gas analysis and/or transcutaneous monitoring in both groups.
  Arms: conventional mechanical ventilation (CMV)

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a complex disorder and remains the most common complication in very preterm infants. Its incidence is increased with gestational age from 95.5% among infants born at 22 weeks' gestation to 22.2% among those born at 29 weeks' gestation. BPD is associated with the increased risks of delayed neurodevelopment and pulmonary impairment. High incidences of BPD and morbidities indicate inadequacy of current management guidelines of BPD.3 Caffeine reduces the development of BPD by lowering the duration of intubation.4 How to further reduce the risk of BPD and the duration of invasive ventilation remain the key focus for neonatologists.

DETAILED DESCRIPTION:
Before 2017, the management guideline of pediatric and adult acute respiratory distress syndrome (ARDS) exclude perinatal triggers-induced ARDS. Moreover, there is insufficient evidence to recommend high-frequency oscillatory ventilation (HFOV) or conventional mechanical ventilation (CMV) as the preferred fist-line therapy in pediatric and adult ARDS. In contrast, HFOV may benefit preterm baboons with acute pulmonary dysfunction-typically due to respiratory distress syndrome (RDS)-by using low tidal volume, supra-physiologically higher respiratory rate, and lower peak inspiratory pressure to enhance oxygenation and gas exchange. The team also reported that use of HFOV is associated with a modest reduction referring to BPD. However, European consensus guideline of RDS only recommend HFOV being a reasonable alternative to CMV when high pressure is needed to achieve adequate lung inflation. Because randomized controlled trials in humans have yielded inconsistent findings.

These differences between animal models-where RDS was induced and treated with surfactant alone-and clinical scenarios, where preterm birth often involved complex etiologies requiring both surfactant and antibiotics for placental insufficiency or intrauterine infection, may be the diagnosis of RDS and ARDS or the mixture of RDS and ARDS. Such findings highlighted the lack of robust evidence for optimizing ventilation strategies in preterm infants born <32 weeks with perinatal ARDS, and the need for well-designed multi-center randomized controlled trials in this high-risk population.

ELIGIBILITY:
Inclusion criteria

1. GA was between 24+0 and 31+6 weeks.
2. Preterm neonates were admitted to NICU within 1 hours after birth, diagnosed with perinatal ARDS using Montreux guidelines and stable supported by CMV.
3. Stabilization for 2 hours before randomization: FiO2 0.40, mean airway pressure (MAP) 10-14 cmH2O, ≤ 40 bpm of respiratory rate, 90%-94% of SpO2, pH > 7.20, PaCO2 60 mmHg, tidal volume of 5 ml/kg and > 35% of hematocrit (these may be evaluated by arterial blood gas analysis).

Exclusion criteria

Neonates were not included if any of the following criteria were met:

1. Parents or guardians' decision not to participate.
2. Major congenital anomalies or chromosomal abnormalities
3. Need for surgery or more than grade 2nd of IVH before randomization.

Ages: 1 Minute to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of bronchopulmonary dysplasia(BPD) | 36 weeks' gestational age
  BPD is defined according to the 2019 diagnostic criteria. For infants discharged before 36 weeks' GA, BPD severity was assessed based on respiratory support at the time of discharge. Infants receiving no supplemental respiratory support were divided into no BPD, those treated with nasal cannula (≤ 2 L/min) as grade 1 BPD, those treated with nasal cannula (> 2 L/min) or noninvasive positive airway pressure as grade 2 BPD and those treated with invasive mechanical ventilation as grade 3 BPD.

SECONDARY OUTCOMES:
duration of invasive ventilation | 36 weeks' gestational age
  duration of invasive ventilation for HFOV or CMV
mortality | 36 weeks' gestational age or before discharge
  the included neonates were diagnosed with death
air leak (pneumothorax and/or pneumomediastinum) occurred | 36 weeks' gestational age or before discharge
  the included neonates were diagnosed with air leak
the incidence of hemodynamically significant patent ductus arteriosus (hsPDA) | 36 weeks' gestational age or before discharge
  the included neonates were diagnosed with hsPDA.
the incidence of retinopathy of prematurity(ROP)> 2nd grades | 36 weeks' gestational age or before discharge
  ROP was categorized according to the International Classification of Retinopathy of Prematurity, revised in 2005
the incidence of necrotizing enterocolitis(NEC)≥2nd stages | 36 weeks' gestational age or before discharge
  the development of NEC, specifically focusing on cases classified as Bell's stage ≥2, according to the modified Bell's staging criteria for NEC.
intraventricular hemorrhage(IVH)>2nd grade | 36 weeks' gestational age or before discharge
  IVH with grades 1-4 were defined by Papile et al

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No